CLINICAL TRIAL: NCT04157920
Title: Impact of Balloon Predilatation Between Self-expanding Valves in All Comers Undergoing TAVI
Brief Title: Impact of Predilatation Between Self-expanding Valves
Acronym: DIRECTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Naval Hospital, Athens (Other); Silesian Centre for Heart Diseases (Other); University General Hospital of Heraklion (Other); Interbalkan Medical Center, Thessaloniki, Greece (Unknown)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Professor, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DIRECT II
Record Dates: First submitted 2019-10-30; First posted 2019-11-08 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Aortic Stenosis
Keywords: Aortic stenosis; DIRECT; ACURATE; TAVI; TAVR; transcatheter; valve
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Intervention Model Description: Patients undergoing TAVR for severe aortic stenosis with two different transcatheter devices. One arm received Medtronic Evolut R/Pro. The other is receiving Boston Scientific ACURATE NEO/TF
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients treated with Medtronic CoreValve/ Evolut R/Pro (Other): TAVI patients treated with Medtronic CoreValve /Evolut R - Evolut PRO Transcatheter Heart Valves, participated in the DIRECT trial
  Interventions: Device: Transcatheter Aortic Valve Implantation with Medtronic CoreValve /Evolut R/Pro
- Patients treated with ACURATE neo/TF (Active Comparator): TAVI patients treated with ACURATE neo/TF Transcatheter Heart Valve recruited prospectively.
  Interventions: Device: Transcatheter Aortic Valve Implantation with ACURATE NEO/TF

INTERVENTIONS:
Device: Transcatheter Aortic Valve Implantation with ACURATE NEO/TF — Transcatheter implantation of the heart valve device ACURATE neo/TF in patients suffering from severe aortic stenosis and are candidates for this operation
  Other Names: Boston Scientific ACURATE neo/TF
  Arms: Patients treated with ACURATE neo/TF
Device: Transcatheter Aortic Valve Implantation with Medtronic CoreValve /Evolut R/Pro — Transcatheter implantation of the heart valve device Medtronic Evolut R/Pro in patients suffering from severe aortic stenosis and are candidates for this operation
  Other Names: Medtronic CoreValve /Evolut R/Pro
  Arms: Patients treated with Medtronic CoreValve/ Evolut R/Pro

SUMMARY:
A Multicenter, prospective, non-randomized, trial evaluating the safety and clinical efficacy of the next-generation, self-expandable Boston Scientific ACURATE NEO/TF Transcatheter Heart Valves, implanted in patients with severe aortic stenosis and the impact of predilatation in comparison with the Medtronic CoreValve EvolutT R/PRO systems from the DIRECT trial.

DETAILED DESCRIPTION:
The aim of the present prospective, multicenter, non-randomized trial is to compare the device success rate and the in-hospital and 30-day safety and echocardiographic clinical outcomes between TAVI with and without predilatation in all comers undergoing implantation of self-expanding valves. Primary endpoint will be device success rate as defined by the VARC-2 criteria. Secondary endpoints involve the composite endpoint of early safety at 30 days, according to the VARC-2 definitions, specifically all cause mortality, cardiovascular mortality, stroke, acute kidney injury, life-threatening or disabling bleeding, major vascular complication, as well as the echocardiographic outcomes and valve performance as designated by the VARC-2 definitions at 30 days. VARC-1 and VARC-3 device success rates will be estimated as well.

Study type: Observational

Estimated Enrollment: 75 patients

Allocation: Non - randomized, all comers

Primary Purpose: Treatment

Observational Model: Case-Control

Condition or disease: Aortic valve stenosis

Intervention/Treatment: Device: Boston Scientific ACURATE neoTM transfemoral TAVI system

Time Perspective: Prospective

Participating centers: Hippokration Hospital (Athens, Greece), Silesian Center for Heart Diseases (Zabrze, Poland), Athens Naval Hospital (Athens, Greece). It is possible that the number of the participating center may change.

Methods: Patients treated with the Boston Scientific ACURATE NEO/TF system will be prospectively. All patients will be followed for at least 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patient with severe symptomatic aortic stenosis defined by a mean aortic gradient > 40 mmHg or peak jet velocity > 4.0 m/s or an aortic valve area (AVA) < 1cm2 or AVA indexed to body surface area (BSA) of <0.6 cm2/m2
* Patient is symptomatic (heart failure with New York Heart Association (NYHA) Functional Class > I, angina or syncope)
* Patients are considered at high risk for mortality with conventional surgical aortic valve replacement as assessed by a Heart Team consisting of a cardiologist and surgeon or as confirmed by a logistic EuroSCORE I ≥ 20% and / or EuroSCORE II ≥ 7% STS score ≥ 8% OR
* Over 80 years old OR
* Over 65 years old with 1 or 2 (but not more than two) from the following criteria:

Liver cirrhosis (Class A or B). Pulmonary insufficiency: VMS<1 liter. Previous heart surgery (CABG, vascular surgery). Porcelain aorta. Pulmonary artery systolic pressure >60 mmHg and high risk for heart surgery. Relapsing pulmonary embolism. Right ventricular insufficiency. Thoracic wall injuries that contraindicate an open heart surgery. History of radiation therapy of the mediastinum. Connective tissue disease that contraindicates an open heart surgery. Frailty/cachexia.

* Aortic valve diameter of ≥20mm and ≤2 9mm as measured by echo.
* Ascending aorta diameter ≤ 43 mm at the sinotubular junction.
* Arterial aorto-iliac-femoral axis suitable for transfemoral access as assessed by conventional angiography and/or multi-detector computed tomographic angiography (access vessel diameter ≥ 6mm)
* Patient understands the purpose, the potential risks as well as benefits of the trial and is willing to participate in all parts of the follow-up
* Patient has given written consent to participate in the trial

Exclusion Criteria:

* A known hypersensitivity or contraindication to any of the following which cannot be adequately pre-medicated: aspirin or heparin and bivalirudin, ticlodipine and clopidogrel, nitinol (titanium or nickel), contrast media
* Ongoing sepsis, including active endocarditis.
* Any percutaneous coronary or peripheral interventional procedure with a bare metal or drug eluting stent performed within 30 days prior to Heart Team assessment.
* Echocardiographic evidence of LV or LA thrombus.
* Mitral or tricuspid valve insufficiency (> grade II).
* Previous aortic valve replacement (mechanical or bioprosthetic).
* Recent (within 6 months of Heart Team assessment) cerebrovascular accident (CVA) or transient ischemic attack (TIA).
* Patients with:

Femoral, iliac or aortic vascular disease (stenosis etc) that precludes the insertion of a transcatheter sheath.

OR Symptomatic carotid or vertebral artery disease (> 70% stenosis).

* The patient has a bleeding diathesis, coagulopathy or denies blood transfusion.
* Estimated life expectancy of less than 12 months due to associated non-cardiac co-morbid conditions.
* Creatinine clearance < 20 ml/min.
* Active gastritis or gastrointestinal ulcer.
* Pregnancy.
* Severe left ventricular dysfunction with left ventricular ejection fraction (LVEF) < 20%.
* Unicuspid aortic valve.
* Mixed aortic valve disease (aortic stenosis and aortic regurgitation> 2+).
* Liver failure (Child-Pugh class C).
* Severe dementia (resulting in either inability to provide informed consent for the study/procedure, prevents independent lifestyle outside of a chronic care facility, or will fundamentally complicate rehabilitation from the procedure or compliance with follow-up visits).
* Extreme aortic valve calcification and calcific asymmetry (Agatston score: grade 4 AgS>5000 AU).
* Aortic valve area of < 0.4 cm2.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2019-09-17 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Device success | 30 days
  ACURATE NEO/TF device implantation success rates, as designated by the VARC-2 criteria

SECONDARY OUTCOMES:
All cause Mortality | 30 days
  Death teates during the hospitalization of the patient, as designated by the VARC-2 criteria
All stroke | 30 days
  Cerebrovascular accident rates during and after the hospitalization of the patient, as designated by the VARC-2 criteria
New pacemaker implantation | 30 days
  New pacemaker implantation rates during and after the hospitalization of the patient, as designated by the VARC-2 criteria
Major Vascular complications | 30 days
  Vascular complications rates during and after the hospitalization of the patient, as designated by the VARC-2 criteria
Echocardiographic endpoint | 30 days
  Echocardiographic endpoint (Post TAVI aortic valve area in cm2)
Post-dilatation | 30 days
  Post-dilatation rates
Major Bleeding | 30 days
  Major bleeding during and after the hospitalization of the patient, as designated by the VARC-2 criteria
Acute kidney injury stage 2 or 3 | 30 days
  AKI stage 2 or 3 during and after the hospitalization of the patient, as designated by the VARC-2 criteria
Device success | 30 days
  ACURATE NEO/TF device implantation success rates, as designated by the VARC-1 and VARC-3 criteria

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos P Toutouzas, Professor, Study Director — Professor of Cardiology
Locations (1):
- Hippocration Hospital First Department of Cardiology, University of Athens, Medical School, Athens, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arora S, Strassle PD, Ramm CJ, Rhodes JA, Vaidya SR, Caranasos TG, Vavalle JP. Transcatheter Versus Surgical Aortic Valve Replacement in Patients With Lower Surgical Risk Scores: A Systematic Review and Meta-Analysis of Early Outcomes. Heart Lung Circ. 2017 Aug;26(8):840-845. doi: 10.1016/j.hlc.2016.12.003. Epub 2017 Jan 24. PMID 28169084
- [Background] Adams HSL, Ashokkumar S, Newcomb A, MacIsaac AI, Whitbourn RJ, Palmer S. Contemporary review of severe aortic stenosis. Intern Med J. 2019 Mar;49(3):297-305. doi: 10.1111/imj.14071. PMID 30091235
- [Background] Saikrishnan N, Kumar G, Sawaya FJ, Lerakis S, Yoganathan AP. Accurate assessment of aortic stenosis: a review of diagnostic modalities and hemodynamics. Circulation. 2014 Jan 14;129(2):244-53. doi: 10.1161/CIRCULATIONAHA.113.002310. No abstract available. PMID 24421359
- [Background] 4. Piérard L. Transcatheter aortic valve implantation: indications. E-Journal of Cardiology Practice [Internet]. 2016 5 May 2019 [cited 2019 5 May 2019]; Volume 14 Available from: https://www.escardio.org/Journals/E-Journal-of-Cardiology-Practice/Volume-14/transcatheter-aortic-valve-implantation-indications
- [Background] Mollmann H, Diemert P, Grube E, Baldus S, Kempfert J, Abizaid A. Symetis ACURATE TF aortic bioprosthesis. EuroIntervention. 2013 Sep 10;9 Suppl:S107-10. doi: 10.4244/EIJV9SSA22. No abstract available. PMID 24025946
- [Background] Manoharan G, Walton AS, Brecker SJ, Pasupati S, Blackman DJ, Qiao H, Meredith IT. Treatment of Symptomatic Severe Aortic Stenosis With a Novel Resheathable Supra-Annular Self-Expanding Transcatheter Aortic Valve System. JACC Cardiovasc Interv. 2015 Aug 24;8(10):1359-1367. doi: 10.1016/j.jcin.2015.05.015. PMID 26315740
- [Background] Forrest JK, Mangi AA, Popma JJ, Khabbaz K, Reardon MJ, Kleiman NS, Yakubov SJ, Watson D, Kodali S, George I, Tadros P, Zorn GL 3rd, Brown J, Kipperman R, Saul S, Qiao H, Oh JK, Williams MR. Early Outcomes With the Evolut PRO Repositionable Self-Expanding Transcatheter Aortic Valve With Pericardial Wrap. JACC Cardiovasc Interv. 2018 Jan 22;11(2):160-168. doi: 10.1016/j.jcin.2017.10.014. PMID 29348010
- [Background] Toutouzas K, Benetos G, Voudris V, Drakopoulou M, Stathogiannis K, Latsios G, Synetos A, Antonopoulos A, Kosmas E, Iakovou I, Katsimagklis G, Mastrokostopoulos A, Moraitis S, Zeniou V, Danenberg H, Vavuranakis M, Tousoulis D. Pre-Dilatation Versus No Pre-Dilatation for Implantation of a Self-Expanding Valve in All Comers Undergoing TAVR: The DIRECT Trial. JACC Cardiovasc Interv. 2019 Apr 22;12(8):767-777. doi: 10.1016/j.jcin.2019.02.005. Epub 2019 Mar 27. PMID 30928442
- [Background] Pagnesi M, Kim WK, Conradi L, Barbanti M, Stefanini GG, Zeus T, Pilgrim T, Schofer J, Zweiker D, Testa L, Taramasso M, Hildick-Smith D, Abizaid A, Wolf A, Van Mieghem NM, Sedaghat A, Wohrle J, Khogali S, Van der Heyden JAS, Webb JG, Estevez-Loureiro R, Mylotte D, MacCarthy P, Brugaletta S, Hamm CW, Bhadra OD, Schafer U, Costa G, Tamburino C, Cannata F, Reimers B, Veulemans V, Asami M, Windecker S, Eitan A, Schmidt A, Bianchi G, Bedogni F, Saccocci M, Maisano F, Alsanjari O, Siqueira D, Jensen CJ, Naber CK, Ziviello F, Sinning JM, Seeger J, Rottbauer W, Brouwer J, Alenezi A, Wood DA, Tzalamouras V, Regueiro A, Colombo A, Latib A. Transcatheter Aortic Valve Replacement With Next-Generation Self-Expanding Devices: A Multicenter, Retrospective, Propensity-Matched Comparison of Evolut PRO Versus Acurate neo Transcatheter Heart Valves. JACC Cardiovasc Interv. 2019 Mar 11;12(5):433-443. doi: 10.1016/j.jcin.2018.11.036. PMID 30846081